CLINICAL TRIAL: NCT03411564
Title: Lights, Camera and Action Against Dating Violence!
Brief Title: Lights, Camera and Action Against Dating Violence (Lights4Violence)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Carmen Vives-Cases, Principal Investigator, University of Alicante
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 776905
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Violence in Adolescence
Keywords: dating violence; health promotion; educational intervention; health assets; participation action research

STUDY DESIGN:
Intervention Model Description: Longitudinal quasi-experimental educational intervention study. The evaluation will be carried out using an on-line questionnaire distributed to an intervention and a control groups at two time periods: before starting the program (Baseline, time 0 or T0), after finishing the study - including the dissemination phase - (time 1 or T1). In addition, a process evaluation will be carried out with the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Students enrolled in one or two targeted secondary schools in each city who are going to receive the intervention (workshop)
  Interventions: Other: Filming Together to See Ourselves in a New 'Present'
- Grup 0 (No Intervention): Students from other centers with similar socioeconomic characteristics (relating to social characteristics and school location) to the centers.

INTERVENTIONS:
Other: Filming Together to See Ourselves in a New 'Present' — PHASE 0. PRIOR TRAINING 1) Promoting protective assets related to violence together. 10-hour training session with 10-15 secondary school teachers; 2) Identifying our own protective assets against violence. This training activity will be addressed to targeted students. The activity will be carried out in four sessions of 1 hour in duration.
  PHASE 1.PRE-PRODUCTION. 1) Participant activity on building story arguments; and 2) Construction of a technical and literary guide to the video capsules.
  PHASE 2: PRODUCTION.- 1) Rehearsal of the script developed by each group; 2) Preparation and selection of environment, wardrobe and characterization of the roles and, 3) Filming of the video capsules.
  PHASE 3: POST-PRODUCTION.- This phase consists of putting together the short film using the various video capsules.
  PHASE 4: DISSEMINATION. A short film exhibition to provide a space where participants can present their video capsules and briefly explain the production process.
  Arms: Group 1

SUMMARY:
Lights4Violence aims to promote adolescents' capabilities to improve their intimate relationships with peers through different participation approach activities. In order to do that, it is planned to perform a longitudinal quasi-experimental educational intervention study with a quantitative evaluation in 5 different cities: Alicante (Spain), Cardiff (UK), Porto (Portugal), Iasi (Romania) and Lublin (Poland) between 2018 and 2019.

DETAILED DESCRIPTION:
DESIGN: Longitudinal quasi-experimental educational intervention study with a quantitative evaluation.

PILOT STUDY (June - July of 2018): Prior to the implementation of the program in the whole sample, an evaluation pilot study will be carried out with a minimum of 20 adolescents (10 boys and 10 girls) who are finishing the same grade as those who will later receive the intervention in August-September 2018. This pilot study focuses on:

* Determining the competencies and capacities of the participants to carry out the on-line questionnaire.
* Calculating the time it takes the students to complete the questionnaire
* Carrying out an internal validation of the questionnaire (that is, are there different responses to similar questions?) among the study population by calculating internal consistency and validity indices.

The obtained results will be shared among the members of the consortium in order to evaluate possible adaptations considered necessary.

PARTICIPANTS: Two groups of students will be assigned either an intervention or control condition, respectively. The intervention group will be composed of boys and girls aged 13 years or more, studying in secondary schools in the city. The control group will be made up of students from other centers with similar socioeconomic characteristics (relating to social characteristics and school location) to the centers. The evaluation survey will be given to a total of 300 students per country, 120 to 150 from the intervention group and 150 from the control group.

The schools selection will be carried out by contacting different secondary education centers from the city as considered appropriate by the members of the research team (non-random sample). The program contents will be presented and the possibility to participate will be offered. The intervention group will be selected from among the students whose centers accept participation in the study. The control group will be made up of students from secondary education centers with social characteristics similar to the centers that will be implement the intervention. The students from the control and the intervention groups will have the same composition in terms of age, sex and academic course. It is recommended that the control and intervention groups belong to different educational centers in order to avoid contamination. It should be mentioned that this is a wait-list control study, that is, those centers that participate in the project as a part of the control group should be offered the possibility of participating in teacher training, access to guides and manuals generated by the project as well as carrying out the intervention in the future (i.e., when the intervention is finished in the intervention group) with Lights4Violence researchers' support if the participants consider it necessary and the research team have the capacity to do it.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 13 to 17 years, studying in the targeted secondary schools in each city.

Exclusion Criteria:

* Students with language barriers

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1555 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Attitudes against sexism | 1-6 months after the intervention
  The Ambivalent Sexism Inventory, a 22-item self-report measure of sexism. Respondents indicate their level of agreement, on a 6-point Likert-type scale, with various statements. It is composed of two sub-scales that may be independently calculated for sub-scale scores or may be averaged for an overall composite sexism score. The first sub-scale is the hostile sexism scale, which is composed of 11 items designed to assess an individual's position on the dimensions of dominative paternalism, competitive gender differentiation, and heterosexual hostility, as previously defined. The second sub-scale is the benevolent sexism scale, which is composed of 11 items that aim to assess an individual's position on the dimensions of protective paternalism, complementary gender differentiation, and heterosexual intimacy.
Level of Aggression | 1-6 months after the intervention
  Aggression Questionnaire-Refined measures four aspects of aggression: Physical Aggression and Verbal Aggression, which involve hurting or harming others and represent the instrumental or motor component of behavior; Hostility, which consists of feelings of ill-will and injustice and represents the cognitive component of behavior; and Anger, which involves physiological arousal and preparation for aggression and represents the emotional or affective component of behavior.
Intolerance towards intimate partner violence | 1-6 months after the intervention
  The Maudsley Violence Questionnaire measures a range of cognitions, relating to violent behavior, drawn from clinical and theoretical perspectives. This measure integrates justification of violence in response to threatened self-esteem and the legitimization of violence as central elements. Participants are asked to rate as True or False a series of statements. The scale is comprised of two factors: 'machismo' (42 items) and 'acceptance of violence' (14 items).

SECONDARY OUTCOMES:
Problem Solving capacity | 1-6 months after the intervention
  The Social Problem-Solving Inventory-Revised Scale is scale of 25 items. Items are answered in a 5-point Likert-type scale, from "this is not true" to "extremely true". Items are distributed in five sub-scales (5 items in each subscale) that evaluate functional and dysfunctional aspects of the ability to problem solve. The functional dimension is evaluated through two sub-scales: Positive Problem Orientation and Rational Problem Resolution; while the dysfunctional dimension is evaluated through the sub-scales Negative Problem Orientation, Avoidance Style and Impulsivity/Carelessness Style. These five dimensions allow obtaining a total score that corresponds to a general estimation of the ability to solve problems, in addition to the average scores in each of the dimensions.
Interpersonal reactivity | 1-6 months after the intervention
  Interpersonal Reactivity Index structure to be made up of four independent dimensions of seven items each: a) Fantasy, which denotes the tendency of the subjects to identify with fictitious subjects such as characters from books and movies, b) Perspective taking, which contains items that reflect the tendency or ability of the subjects to adopt the perspective or point of view of other people, c) Empathetic concerns, which contains items that evaluate the subject's tendencies to experience sensations of compassion and concern towards others, and d) Personal distress, which includes items that indicate that subjects experience feelings of discomfort and anxiety when witnessing the negative experiences of others. Respondents rate how well several statements describe them, on a 5-point Likert type scale from "does not describe me well" to "describes me very well".
Self-esteem | 1-6 months after the intervention
  Rosenberg Self-Esteem Scale is a 10-item scale that measures global self-worth by assessing both positive and negative feelings about the self. The scale is believed to be unidimensional. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree.
Assertiveness | 1-6 months after the intervention
  Measured by the Assertive Interpersonal Schema Questionnaire with 21 items, assesses four dimensions that refer to external emotional support (5 items), practical personal ability (4 items), interpersonal management (8 items) and affective personal ability (4 items). Items are rated on a 1 (completely false) to 5 (completely true) Likert-type scale. Scores on the questionnaire higher than the average in each of the dimensions indicate good personal adjustment and adequate capacity for assertiveness.

OTHER OUTCOMES:
Subjective happiness | 1-6 months after the intervention
  The Subjective Happiness Scale is a global measure of subjective happiness that evaluates wellbeing as a global psychological phenomenon, considering the definition of happiness from the perspective of the respondent. It consists of four items with Likert-type responses with 7 options. Scores are the total number of items divided by the sum of the scores obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Vives-Cases, Dr, Principal Investigator — University of Alicante
Locations (1):
- University of Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanz-Barbero B, Ayala A, Ieracitano F, Rodriguez-Blazquez C, Bowes N, De Claire K, Mocanu V, Anton-Paduraru DT, Sanchez-SanSegundo M, Albaladejo-Blazquez N, das Neves ASA, da Silva Queiros AS, Jankowiak B, Waszynska K, Vives-Cases C. Effect of the Lights4Violence intervention on the sexism of adolescents in European countries. BMC Public Health. 2022 Mar 19;22(1):547. doi: 10.1186/s12889-022-12925-3. PMID 35305589
- [Derived] Vives-Cases C, Sanz-Barbero B, Ayala A, Perez-Martinez V, Sanchez-SanSegundo M, Jaskulska S, Antunes das Neves AS, Forjaz MJ, Pyzalski J, Bowes N, Costa D, Waszynska K, Jankowiak B, Mocanu V, Davo-Blanes MC. Dating Violence Victimization among Adolescents in Europe: Baseline Results from the Lights4Violence Project. Int J Environ Res Public Health. 2021 Feb 3;18(4):1414. doi: 10.3390/ijerph18041414. PMID 33546373
- [Derived] Vives-Cases C, Davo-Blanes MC, Ferrer-Cascales R, Sanz-Barbero B, Albaladejo-Blazquez N, Sanchez-San Segundo M, Lillo-Crespo M, Bowes N, Neves S, Mocanu V, Carausu EM, Pyzalski J, Forjaz MJ, Chmura-Rutkowska I, Vieira CP, Corradi C. Lights4Violence: a quasi-experimental educational intervention in six European countries to promote positive relationships among adolescents. BMC Public Health. 2019 Apr 8;19(1):389. doi: 10.1186/s12889-019-6726-0. PMID 30961558